CLINICAL TRIAL: NCT04342559
Title: Evaluation Of Acceptability, Under Use in Real Conditions Of Two Vaginal Moistures ( 06260308 ) Indicated for Women With Vaginal Drying
Brief Title: Acceptability, Under Use in Real Conditions Of Two Vaginal Moistures Indicated for Women With Vaginal Drying
Acronym: PRV01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AllSEUGEPpHFL06260307080418
Record Dates: First submitted 2020-04-06; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Vaginal Dryness
Keywords: vaginal hydration

STUDY DESIGN:
Intervention Model Description: Open, non-comparative clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Belamy with sinodor Vaginal Moisturizer with Odor Neutralizer - code: 062603-07
  Participants will be instructed on how to use it as follows:
  Guidance The product has individual pre-filled applicators for single use and disposable after use. The applicator has an anatomical shape, in order to facilitate use, avoiding discomfort during application.
  A single application should be performed every 3 days (72 hours). I use it at night, before going to bed, before going to sleep.
  Interventions: Other: Belamy (vaginal moisturizer)
- Group II (Experimental): Belamy without sinodor Vaginal Moisturizer without Odor Neutralizer - code: 062603-08
  Participants will be instructed on how to use it as follows:
  Guidance The product has individual pre-filled applicators for single use and disposable after use. The applicator has an anatomical shape, in order to facilitate use, avoiding discomfort during application.
  A single application should be performed every 3 days (72 hours). I use it at night, before going to bed, before going to sleep.
  Interventions: Other: Belamy (vaginal moisturizer)

INTERVENTIONS:
Other: Belamy (vaginal moisturizer) — The conformity of the product use by the research participants will be verified through the filling of the product use diary by the research participants and also by the accounting of the tubes not used in T22.
  Interdiction and Restriction
  * Keep the test product tightly closed, protected from heat, moisture and out of the reach of children;
  * Do not apply any other product to the genital area. Only the use of soap normally used for hygiene will be allowed;
  * Do not change genital / vaginal hygiene habits;
  * Not having sexual intercourse in the 48 hours (2 days) before the research visits;
  * Do not perform a hygienic shower in the genital region within 24 hours (1 day) prior to the research visits;
  * Do not perform gynecological / intimate showers during the study period

SUMMARY:
The studies carried out to evaluate the safety and efficacy of products aimed at the intimate area of women aim to confirm the absence of risk associated with its use, identify possible feelings of discomfort and / or clinical signs resulting from the use of the product and evaluate the benefits provided by the use of the product such as, gynecologically tested, clinically tested, hydration for 72 hours, hydration, does not drip or drip little, feeling of natural hydration, control of natural vaginal odor, preserves vaginal pH, does not promote irritation, use vaginal topic, feeling of comfort, relief from dryness, easy use of the applicator, the applicator does not cause discomfort during application, preferably use at night, does not change the vaginal flora, reduces pain and discomfort during or shortly after sexual intercourse, does not promote discomfort during or shortly after intercourse, reduction of vaginal bleeding during or right after sexual intercourse, if there is a small amount left in the applicator, the treatment is not compromised.

The research will be carried out with two new products for use in the internal intimate region in up to 74 research participants (up to 37 participants per product - each group of 37 will use one of the products), which meet the required inclusion and exclusion criteria. At the end of the treatment, the analysis must contain a minimum number of 30 participants per product. Participants will use the test products for 22 (+ 2) days and will be evaluated and monitored throughout the study by a gynecologist to verify the effectiveness of the products and possible adverse events. In addition, a profile questionnaire will be applied at the beginning of the study (T0 - day 1) and at the end of the study, the perceived efficacy questionnaire (T22), to assess signs and symptoms of the efficacy and safety of the product used.

DETAILED DESCRIPTION:
Moisturizers are used in chronic maintenance, replacing normal vaginal sections.

Vaginal moisturizers rehydrate the mucosal tissue and are absorbed by the skin, adhering to the vaginal lining, thus mimicking natural vaginal secretions. The use of vaginal moisturizers is intended to allow dryness / atrophy, vaginitis / non-hormonal vaginal atrophy and is regularly harmful or once every 2-3 days. The frequency of use is directly proportional to the severity of the atrophy (for example, the more severe the atrophy, the more frequent the application is), the effects of the moisturizer are more prolonged and the effects of the lubricant, lasting 2 to 3 days.

MOD_PRO_CEP Rev. 03 All-SE-UG-EP-pH-FL-062603-07 / 08-04-18-PRV01 Vaginal moisturizers use this longer to change the content of the endothelium fluid, capture the vaginal pH and thus maintain vaginal hydration and acidity. Therefore, they are particularly beneficial, not only for women with VVA / GSM symptoms that cause pain during intercourse, but also for women who are not currently sexually active, but experience discomfort on a daily basis. Since vaginal moisturizers are used to moisturize the mucosa, most contain water. For the water to stick to the mucosa, it also contains vegetable or synthetic polymers. In addition, they can use a wide variety of other excipients to provide adequate viscosity, to buffer or pH and for conservation; these additional ingredients (some synthetic polymers) affect the pH and osmolality of the moisturizer.

The products to be tested in this study are two vaginal moisturizers. These are two new products from the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy research participants with an active sex life;
* Skin and intact mucosa in the test region;
* Agreement to adhere to the study's procedures and requirements and to attend the institute on the day (s) and time (s) determined for the assessments;
* Ability to consent to their participation in the study;
* Female research participants;
* Menopausal participants of any age;
* Participants who complain of vaginal dryness, classified at least as mild, and who present at least one of the following symptoms, in addition to vaginal dryness, also classified at least as mild (pain during or shortly after intercourse or discomfort during or soon after sexual intercourse).

Exclusion Criteria:

* Have used moisturizing creams and / or vaginal lubricants 05 days before the initial study visit;
* Vaginal pathology in the product application area;
* Have had sex less than 48 hours before the visit;
* Have been diagnosed with urogenital or vaginal infection in the last 30 days;
* Have used topical or systemic antibiotics, antifungals, hormone-based creams or treatment for vaginal atrophy in the last six weeks;
* Immune failure;
* Current use of the following medications for topical or systemic use: corticosteroids, immunosuppressants and antihistamines and in the last 7 days;
* History of reaction to the category of the product tested;
* Present vaginal bleeding on the day of visits;
* Other diseases or medications that may directly interfere with the study result or endanger the health of the research participant, at the discretion of the investigator.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Intensity of clinical signs (Visual gynecological examination) | day 1
  Visual examination of the vulva, vagina and cervix using a speculum. Objective vaginal signs will be described, such as: inflammation, edema, presence of abrasions and presence of deepithelialization of the vaginal mucosa in the initial (T0 - Day 1).Each clinical sign will be classified using a scale from 0 to 3 from the best to the worst scenario (0 - Absent, 1 - Mild, 2 - Moderate or 3 - Intense).
Intensity of clinical signs (Visual gynecological examination) | day 22
  Visual examination of the vulva, vagina and cervix using a speculum. Objective vaginal signs will be described, such as: inflammation, edema, presence of abrasions and presence of deepithelialization of the vaginal mucosa in the final (T22- Day 22).Each clinical sign will be classified using a scale from 0 to 3 from the best to the worst scenario (0 - Absent, 1 - Mild, 2 - Moderate or 3 - Intense).
Vaginal pH measurements | day 1
  Before using the product (T0 - day 1), the vaginal pH will be evaluated, with the aid of a speculum, using colorimetric pH measuring tapes, with a gradual scale of 2 to 9.
  The tapes will be applied in contact with the right lateral vaginal wall, without touching the cervix or cervical mucus, due to the pH difference. The cervix, as well as the cervical mucus, have a pH more alkaline than the vagina, and may interfere with the result that will be evaluated by colorimetric approximation using the standard template
Vaginal pH measurements | day 22
  Before using the product after 22 + 2 days (T22), the vaginal pH will be evaluated, with the aid of a speculum, using colorimetric pH measuring tapes, with a gradual scale of 2 to 9.
  The tapes will be applied in contact with the right lateral vaginal wall, without touching the cervix or cervical mucus, due to the pH difference. The cervix, as well as the cervical mucus, have a pH more alkaline than the vagina, and may interfere with the result that will be evaluated by colorimetric approximation using the standard template
Bacterioscopic collection | days 1 and 22
  Before using the product (T0 - day 1) and after 22 + 2 days (T22), the bacterioscopic collection of vaginal secretion will be performed to quantify the microorganisms present in it in order to assess the non-interference of the use of the product in the flora vaginal.
  The collection of vaginal material from the participants will be performed by a gynecologist with the insertion of a speculum in the vagina. The excess cervical mucus will be removed with the aid of MOD_PRO_CEP Rev. 03 All-SE-UG-EP-pH-FL-062603-07 / 08-04-18-PRV01 cotton swab. Then, the swabs indicated for collection will be inserted and rotated for a few seconds on the bottom of the vaginal sac.The swabs containing the samples will be immediately placed in sterile test tubes and sent to the laboratory for microbiological analysis.
Visual assessment of product accumulation in the mucosa | after 72 hours
  Visual assessment of accumulation of product adhered to the mucosa will be performed after 72 hours or more, considering the study window (+2 days), without using the product (T22):
  0: Absent
  1. Little buildup
  2. Moderate accumulation
  3. Intense accumulation
Vaginal Health Index | after 72 hours
  Classification by the gynecologist of the parameters present in the vaginal health score (Vaginal Health Index) before and after using the product (T0 - day 1 and T22 + 2 days), as shown below.
  During the specular examination, a vaginal health index will be evaluated by the gynecologist, with scores from 1 to 5. A lower score corresponds to greater urogenital atrophy (worse outcome)
Teste de Contato (patch test) | up to 22 day
  If, during the research, any participant has an adverse reaction such as contact dermatitis, they will be subjected to epicutaneous tests. The evaluation scale to be used will be the scale recommended by the International Contact Dermatitis Investigator Group - ICDRG -

SECONDARY OUTCOMES:
Evaluation of Effectiveness Perceived by Research Participants | day 1
  Before using the product (T0 - day 1) of use, the research participants will be instructed to self-assess themselves through of questionnaires.A point scale will be used, using a numerical scale (0 to 4) to assess this perception (0 - worse outcome to 4-better outcome)
Evaluation of Effectiveness Perceived by Research Participants | day 22
  Before using the product after 22 + 2 days (T22) of use, or only after using the product (T22), the research participants will be instructed to self-assess themselves through of questionnaires.A point scale will be used, using a numerical scale (0 to 4) to assess this perception (0 - worse outcome to 4-better outcome)
Rate of Gynecological Adverse Reactions | up to 22 day
  All reactions will be classified according to their intensity, according to the classification below (From best -mild to worst scenario -intense):
  Mild: Awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with the participant's usual functions or normal daily activities.
  Moderate: enough discomfort present to cause interference with a part of the participant's usual functions or normal daily activities.
  Intense: Extreme difficulty, causing significant damage to functioning or disability; significantly interferes with the participant's usual functions; prevents normal daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusto Theodoro de Figueiredo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No